CLINICAL TRIAL: NCT00001486
Title: A Neurobiological Investigation of Patients With Schizophrenia Spectrum Disorders and Their Siblings
Brief Title: Genetic Study of Schizophrenia
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950150; 95-M-0150
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01-14

CONDITIONS: Schizoaffective Disorder; Schizophrenia
Keywords: Negative Symptoms; Brain Scans; Hallucinations; Delusions; Psychosis and Schizophrenia; Natural History
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Hallucinations; Delusions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal Controls: Male and female adult healthy volunteers
- Parents: Parents of Probands and siblings for the purposes of DNA collection
- Probands: Adult Subjects with Schizophrenia Spectrum Disorders
- Siblings: Adult siblings of Probands

SUMMARY:
This large ongoing study at NIMH investigates the neurobiology of schizophrenia by identifying susceptibility genes, evaluating their impact on brain function to better understand how to treat and prevent this illness....

DETAILED DESCRIPTION:
Objective: Schizophrenia is a complex genetic disorder which likely involves many genes each producing a slight increase in risk. Finding weak-acting genes in complex genetic disorders has been challenging and will likely require a number of approaches and large clinical samples. Several strategies have emerged recently that appear to markedly improve the power of genetic studies for detecting such genes. These include using association (rather than linkage) and using intermediate phenotypes in addition to DMS-IV diagnosis.

Study Population: We propose to take advantage of these techniques by studying quantitative traits related to schizophrenia in patients, siblings, and controls.

Design: We will employ an association design, rather than linkage. Traits will include quantifiable neurobiological variables that have been implicated previously as possible phenotypes related to schizophrenia. These include tests of attention and cognition.

Outcome Measure: We will use several statistical methods to show that specific genetic polymorphisms affect these phenotypes, including case control and family based association studies.

ELIGIBILITY:
* INCLUSION/EXCLUSION CRITERIA:

Inclusion criteria for Siblings (probands and unaffected siblings):

* Probands must have a DSM IV-R diagnosis of schizophrenia,schizoaffective disorder, psychosis N.O.S. or schizophreniform disorder.
* Probands and Siblings must be between the ages of 18 and 55
* Probands and Siblings must be free of major medical illnesses, but may have controlled hypertension, thyroid disease, or diabetes.
* Probands and Siblings must have the cognitive ability to consent for themselves. Those who are judged to have the cognitive ability to consent for themselves at the time of participation, but do not have the legal capacity to consent for themselves may participate if the legal guardian /Legal authorized representative (LAR) provides consent by signing the informed consent form.
* Fluency in English is required.

Exclusion Criteria for Siblings (probands and unaffected siblings):

* Seizure disorder, mental retardation, organic brain damage or other neurological disease.
* History of any (excepting nicotine-related) DSM5-defined moderate to severe substance use disorder (or DSM-IV-defined substance dependence).
* Cumulative lifetime history of any (excepting nicotine-related) DSM5-defined mild substance use disorder (or any DSM-IV-defined substance abuse), either in excess of 5 years total or not in remission for at least 6 months.
* Head trauma with loss of consciousness over 5 minutes from all but genetic sampling.
* Chemotherapy.
* NIMH employees/staff and their immediate family members will be excluded from the study per NIMH policy

Siblings who do not qualify for the 2-day or 1-day study, may participate in the limited phenotyping arm in which only a psychiatric interview and a blood draw for genetic analysis (SCID-DNA) will be performed, case control analysis or be included as part of a trio (one parent, one sibling, one patient) to study genetic transmission from parents to offsprings.. All parents are eligible for the study.

Inclusion Criteria. Healthy Volunteers/Controls

To be eligible for this research study, healthy volunteers must be:

* Between the ages of 18 and 55
* Fluency in English is required

Healthy Controls Exclusion Criteria:

They will not be eligible if:

* They have history of DSM IV-R psychiatric diagnosis or severe chronic medical illness at the time of the study.
* They have a history of any (excepting nicotine-related) DSM5-defined moderate to severe substance use disorder (or DSM-IV-defined substance dependence).
* They have a cumulative lifetime history of any (excepting nicotine-related) DSM5-defined mild substance use disorder (or any DSM-IV-defined substance abuse), either in excess of 5 years total or not in remission for at least 6 months.
* They may not be eligible for the 2-day or 1-day study if they have a first-degree relative with history of schizophrenia spectrum disorders. However, they may be included in the SCID_DNA or case control analyses.
* Healthy volunteers must be free of learning disabilities.
* NIMH employees/staff and their immediate family members will be excluded from the study per NIMH policy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Probands, healthy controls, siblings, parents
Sampling Method: Probability Sample
Enrollment: 4914 (Actual)
Dates: Start 1995-07-15 (Actual)

PRIMARY OUTCOMES:
Genetic Polymorphisms affect phenotypes | At time of study participation
  genotyping analysis

SECONDARY OUTCOMES:
PANSS, AIMS, GAF | At time of study participation
  PANSS, AIMS, GAF

CONTACTS AND LOCATIONS:
Overall Officials: Karen F Berman, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cloninger CR. Genetic principles and methods in high-risk studies of schizophrenia. Schizophr Bull. 1987;13(3):515-23. doi: 10.1093/schbul/13.3.515. PMID 3306908
- [Background] Cornblatt BA, Keilp JG. Impaired attention, genetics, and the pathophysiology of schizophrenia. Schizophr Bull. 1994;20(1):31-46. doi: 10.1093/schbul/20.1.31. PMID 8197420
- [Background] Holzman PS, Kringlen E, Levy DL, Haberman SJ. Deviant eye tracking in twins discordant for psychosis. A replication. Arch Gen Psychiatry. 1980 Jun;37(6):627-31. doi: 10.1001/archpsyc.1980.01780190025002. PMID 7190001
- [Derived] Kippenhan JS, Gregory MD, Nash T, Kohn P, Mervis CB, Eisenberg DP, Garvey MH, Roe K, Morris CA, Kolachana B, Pani AM, Sorcher L, Berman KF. Dorsal visual stream and LIMK1: hemideletion, haplotype, and enduring effects in children with Williams syndrome. J Neurodev Disord. 2023 Aug 26;15(1):29. doi: 10.1186/s11689-023-09493-x. PMID 37633900
- [Derived] Page SC, Sripathy SR, Farinelli F, Ye Z, Wang Y, Hiler DJ, Pattie EA, Nguyen CV, Tippani M, Moses RL, Chen HY, Tran MN, Eagles NJ, Stolz JM, Catallini JL 2nd, Soudry OR, Dickinson D, Berman KF, Apud JA, Weinberger DR, Martinowich K, Jaffe AE, Straub RE, Maher BJ. Electrophysiological measures from human iPSC-derived neurons are associated with schizophrenia clinical status and predict individual cognitive performance. Proc Natl Acad Sci U S A. 2022 Jan 18;119(3):e2109395119. doi: 10.1073/pnas.2109395119. PMID 35017298
- [Derived] Ursini G, Punzi G, Langworthy BW, Chen Q, Xia K, Cornea EA, Goldman BD, Styner MA, Knickmeyer RC, Gilmore JH, Weinberger DR. Placental genomic risk scores and early neurodevelopmental outcomes. Proc Natl Acad Sci U S A. 2021 Feb 16;118(7):e2019789118. doi: 10.1073/pnas.2019789118. PMID 33558239
- [Derived] Toulopoulou T, Zhang X, Cherny S, Dickinson D, Berman KF, Straub RE, Sham P, Weinberger DR. Polygenic risk score increases schizophrenia liability through cognition-relevant pathways. Brain. 2019 Feb 1;142(2):471-485. doi: 10.1093/brain/awy279. PMID 30535067
- [Derived] Marenco S, Meyer C, van der Veen JW, Zhang Y, Kelly R, Shen J, Weinberger DR, Dickinson D, Berman KF. Role of gamma-amino-butyric acid in the dorsal anterior cingulate in age-associated changes in cognition. Neuropsychopharmacology. 2018 Oct;43(11):2285-2291. doi: 10.1038/s41386-018-0134-5. Epub 2018 Jul 3. PMID 30050047
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1995-M-0150.html